CLINICAL TRIAL: NCT01521117
Title: A Randomized, Double-blind, Placebo Controlled, Crossover Study to Evaluate the Effect of Donepezil on Gait and Balance in Parkinson's Disease
Brief Title: The Effect of Donepezil on Gait and Balance in Parkinson's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Amie Hiller, MD, Principal Investigator, Oregon Health and Science University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: OHSU-7363
Record Dates: First submitted 2012-01-12; First posted 2012-01-30 (Estimated); Results first posted 2021-08-27 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Parkinson's Disease
Keywords: donepezil; parkinson's disease; balance; cholinesterase inhibitor
MeSH Terms: conditions — Parkinson Disease | interventions — Donepezil; Sugars

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Donepezil, Then Placebo (Experimental): Donepezil 5 mg a day for weeks 1 - 3, if tolerated increased to 10 mg a day for weeks 4 - 6. After a washout period of 4 weeks, placebo 5 mg a day for weeks 1 - 3, if tolerated increased to 10 mg a day for weeks 4 - 6.
  Interventions: Drug: Donepezil; Drug: Placebo
- Placebo, Then Donepezil (Experimental): Placebo 5 mg a day for weeks 1 - 3, if tolerated increased to 10 mg a day for weeks 4 - 6.
  After a washout period of 4 weeks, donepezil 5 mg a day for weeks 1 - 3, if tolerated increased to 10 mg a day for weeks 4 - 6.
  Interventions: Drug: Donepezil; Drug: Placebo

INTERVENTIONS:
Drug: Donepezil — Use 1 capsule (5 mg) of donepezil once per day for first 21 days than donepezil 10mg qday for 21 days.
  Other Names: Aricept
Drug: Placebo — Use 1 capsule (5 mg) once per day for first 21 days than 10mg qday for 21 days.
  Other Names: Sugar Pill

SUMMARY:
This study involves Parkinson's disease (PD). Symptoms include slow movement, tremor, and muscle rigidity. Current medications for the treatment of PD do not improve gait and balance difficulties in individuals with PD. Donepezil (study drug) has been found to reduce falls in individuals with PD. The mechanism in which this reduction of falls occurs is unclear. The investigators study will look at what aspects of gait and balance are improved by the study drug. The study drug is not approved to treat PD in the United States or other countries because we do not know enough about it.

DETAILED DESCRIPTION:
Parkinson's disease (PD) is a common neuro-degenerative disease affecting about 2% of the adult population in the United States over the age of 65. Some of the most disabling symptoms of Parkinson's disease are balance and gait dysfunction, leading to falls. These symptoms do not respond to current dopamine directed therapies. Evidence from both pathologic studies and advanced imaging has demonstrated that a cholinergic deficiency in the thalamus and basal ganglia is found in individuals with PD who fall compared to non-fallers. The central acting acetylcholine esterase inhibitor, donepezil, has been demonstrated to decrease falls in individuals with PD. The mechanism by which falls decreased is unknown. Our open label pilot data indicates that donepezil can improve quantitative measures of balance in individuals with PD. Suggesting that improvements in balance in the mechanism by which donepezil reduces falls. Our goal is to determine whether donepezil will:

* Improve quantitative measures of balance in subjects with Parkinson's disease compared to placebo.
* Improve quantitative measures of gait in subjects with Parkinson's disease compared to placebo.
* Improve cognitive measures in non-demented subjects with Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Idiopathic Parkinson's disease, defined by the UK Brain Bank criteria, with a Hoehn and Yahr score of 2 to 4
* Treated with levodopa for at least a year and on a stable antiparkinsonian regimen for at least one month
* Abnormal computerized dynamic posturography (CDP) on screening defined as a composite score below 65 (range 1-100)

Exclusion Criteria:

* Dementia defined by MMSE less than 27
* Other medical conditions other than PD affecting balance or gait as determined by the investigators
* Unable to stand unassisted for 30 minutes
* Current use of an acetylcholinesterase inhibitors or drugs with known anticholinergic properties
* Medical or psychiatric co-morbidities that may interfere with compliance or might place subject in danger as determined by the investigators

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2011-12; Primary Completion 2012-04 (Actual); Study Completion 2012-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Seth Kareus, MD, Principal Investigator — Movement Disorders Program - Parkinson's Center of Oregon - Oregon Health and Science University
Locations (1):
- Parkinson's Center of Oregon - Oregon Health and Science University, Portland, Oregon, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through a large university movement disorders clinic in the Northwest. Inclusion criteria were idiopathic PD, treated with levodopa for at least a year, on a stable antiparkinson regiment for at least one month, abnormal dynamic posturography. Exclusion criteria: dementia (MMSE < 27), another medical condition affecting gait, unable to stand unassisted for 30 minutes, taking a cholinesterase inhibitor or anticholinergic medication.
Groups:
- Donepezil, Then Placebo: Donepezil: Use 1 capsule (5 mg) of donepezil once per day for first 21 days than donepezil 10mg qday for 21 days. After a washout of 4 weeks, Placebo: Use 1 capsule (5 mg) once per day for first 21 days 10mg qday for 21 days.
- Placebo, Then Donepezil: Placebo: Use 1 capsule (5 mg) once per day for first 21 days 10mg qday for 21 days. After a washout of 4 weeks, Donepezil: Use 1 capsule (5 mg) of donepezil once per day for first 21 days than donepezil 10mg qday for 21 days.
Period: First Intervention (6 Weeks)
Arm/Group | Donepezil, Then Placebo | Placebo, Then Donepezil
Started | 10 | 11
Completed | 5 | 8
Not Completed | 5 | 3
Not completed — Adverse Event | 5 | 1
Not completed — Scheduling Issues | 0 | 2
Period: Washout (4 Weeks)
Arm/Group | Donepezil, Then Placebo | Placebo, Then Donepezil
Started | 5 | 8
Completed | 5 | 8
Not Completed | 0 | 0
Period: Second Intervention (6 Weeks)
Arm/Group | Donepezil, Then Placebo | Placebo, Then Donepezil
Started | 5 | 8
Completed | 5 | 5
Not Completed | 0 | 3
Not completed — Adverse Event | 0 | 3

BASELINE CHARACTERISTICS:
Population: Baseline characteristics are reported on all study completers (N = 10).
Groups:
- Total: Total of all study completers.
Arm/Group | Total
Number analyzed (Participants) | 10
Age, Continuous [Mean (Standard Deviation); unit: years] | 70 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 5
Region of Enrollment [Number; unit: participants]
  United States | 10
Unified Parkinson's Disease Rating Scale - Motor Section [Mean (Standard Deviation); unit: units on a scale] — This is the motor subsection of the Unified Parkinson's Disease Rating Scale (UPDRS) and is a commonly used tool to rate the symptoms of Parkinson's disease. Each item on the scale is rated from 0 (normal) to 4 (Can barely perform the task) several motor areas including speech, facial expression, tremor, rigidity, hand movements, agility, posture, and gait. Total score ranges from 0 to 108 with higher values on this scale represent a more severe stage of the disease.
  units on a scale | 24 (7)
Parkinson's Disease Duration (years) [Mean (Standard Deviation); unit: years] — Number of years since self-reported diagnosis (Diagnosis Year - Screening Visit Year).
  years | 10.5 (8)
Mini-Mental Status Exam (MMSE) [Mean (Standard Deviation); unit: units on a scale] — The Mini-Mental Status Exam (MMSE) is a widely used test of cognition the elderly. It includes tests of orientation to time and place, attention, memory, language, recall, complex commands, and visuo-spatial skills. Each item is score 0 (cannot do) to 1 (can do). All items are summed to a total score (Range 0 - 30). Those with scores 25-30 are not impaired, scores 20-25 are mildly impaired and may require some supervisions, scores 10-20 are moderately impaired, and below 10 are severely impaired and are likely to require 24-hour supervision and assistance with activities of daily living.
  units on a scale | 29.2 (0.4)
Trials B-A [Mean (Standard Deviation); unit: seconds] — The Trail Making Test (TMT) consists of two parts (A & B) in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. The test provides information about visual search speed, scanning, speed of processing, and executive functioning. Part A measures processing speed and part B measures executive functioning. The TMT is time to complete each part of the test in seconds. Higher scores indicate greater impairment. Subtracting A from B (Trails B-A) is theorized to provide a relatively pure indicator of executive function.
  seconds | 59 (32)

OUTCOME MEASURES:

1. Primary Outcome: Sensory Organization Test - Composite Score
Description: Balance was measured using the Sensory Organization test (SOT) on the NeuroCom Balance Master Clinical Research System platform (Neurocom International, Inc), which tests sway in 6 conditions, eyes open, eyes closed, and a moving visual surround first with a stable platform then with a moving platform. Center of Pressure (CoP) was calculated from the recordings. Forces and moments were recorded at 100Hz sampling frequency. A change score from the beginning of each treatment phase (placebo or active drug) to the end of the treatment phase. The SOT is scored on an interval scale with the highest possible score of 100 indicating no sway at all. The lowest possible score of 0 indicates the trial was stopped due to an impending fall. Higher scores are indicative of better balance (greater stability).
Time Frame: Change from Day 1 of each treatment phase to Day 42 of each treatment phase
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Donepezil: Donepezil: Use 1 capsule (5 mg) of donepezil once per day for 21 days
- Placebo: Placebo: Use 1 capsule (5 mg) once per day for 21 days
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 10 | 10
score on a scale | 7.7 (21.6) | 0.6 (8.9)

2. Primary Outcome: Sensory Organization Test (SOT) - Condition 4 (Eyes Open, Moving Surround, Stable Platform).
Description: Condition 4 of the Sensory Organization Test. The participants eyes are open as the surround moves and the platform remains stable. A change score from the beginning of each treatment phase (placebo or active drug) to the end of the treatment phase. The SOT is scored on an interval scale with the highest possible score of 100 indicating no sway at all. The lowest possible score of 0 indicates the trial was stopped due to an impending fall. Higher scores are indicative of better balance (greater stability).
Time Frame: Change from Day 1 of each treatment phase to Day 42 of each treatment phase
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 10 | 10
units on a scale | 6.52 (2.99) | -0.89 (2.82)

3. Secondary Outcome: Trails B - A
Description: The Trail Making Test (TMT) consists of two parts (A & B) in which the subject is instructed to connect a set of 25 dots as quickly as possible while still maintaining accuracy. The test provides information about visual search speed, scanning, speed of processing, and executive functioning. Part A measures processing speed and part B measures executive functioning. The TMT is time to complete each part of the test in seconds. Higher scores indicate greater impairment. Subtracting part A from part B (Trails B-A) is theorized to reduce the influence of the working memory and visuo-spatial demands and, therefore, provides a relatively pure indicator of executive function. A change score from the beginning of each treatment phase (placebo or active drug) to the end of the treatment phase.
Time Frame: Change from Day 1 of each treatment phase to Day 42 of each treatment phase
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Donepezil | Placebo
Number analyzed (Participants) | 10 | 10
seconds | 9.4 (95.6) | 1.4 (39.9)

ADVERSE EVENTS:
Groups:
- Donepezil: Donepezil: Use 1 capsule (5 mg) of donepezil once per day for first 21 days than donepezil 10mg qday for 21 days in either the first or last 6 weeks of the study.
- Placebo: Placebo: Use 1 capsule (5 mg) once per day for first 21 days 10mg qday for 21 days in either the first or last 6 weeks of the study.
Arm/Group | Donepezil | Placebo
All-Cause Mortality (participants affected / at risk) | 0/18 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/18 | 0/16
Other Adverse Events (participants affected / at risk) | 6/18 | 1/16
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Donepezil (N=18) | Placebo (N=16)
Gastrointestinal (Gastrointestinal disorders) | 4 (7) | 0 (0) — Nausea, Diarrhea, Vomiting, or gastrointestinal discomfort
Worsening Parkinsonism (Nervous system disorders) | 1 (1) | 0 (0) — Worsening freezing and balance
Possible Transient ischemic attacks (Nervous system disorders) | 0 (0) | 1 (1)
Fall (General disorders) | 2 (2) | 0 (0) — leading to hospitalization

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes